CLINICAL TRIAL: NCT03519984
Title: A Phase I Dose Escalation Study With Expansion to Evaluate the Safety of SEPHB4-HSA in Combination With Cytarabine or Liposomal Vincristine in Patients With Relapsed or Refractory Acute Leukemia
Brief Title: EphB4-HSA Fusion Protein and Cytarabine /or Liposomal Vincristine in Patients With Recurrent or Refractory Acute Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study drug supply issue
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Vasgene Therapeutics, Inc (Industry); Whittier Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9L-17-15; NCI-2018-00680 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9L-17-15 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2018-04-26; First posted 2018-05-09 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Blasts 5 Percent or More of Bone Marrow Nucleated Cells; Myelodysplastic/Myeloproliferative Neoplasm; Philadelphia Chromosome Positive; Recurrent Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Refractory Acute Lymphoblastic Leukemia; Refractory Acute Myeloid Leukemia; Refractory Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Secondary Acute Myeloid Leukemia; T Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Myelodysplastic-Myeloproliferative Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cytarabine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (sEPHB4-HSA, cytarabine) (Experimental): Participants receive recombinant EphB4-HSA fusion protein IV over 60 minutes on days 1, 8, 15, and 22 and cytarabine IV over 4 hours on days 1-5. Treatment repeats every 28 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cytarabine; Other: Laboratory Biomarker Analysis; Biological: Recombinant EphB4-HSA Fusion Protein
- Arm B (sEPHB4-HSA, vincristine liposomal) (Experimental): Participants receive recombinant EphB4-HSA fusion protein IV over 60 minutes on days 1, 8, 15, and 22 and vincristine liposomal IV over 60 minutes on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Recombinant EphB4-HSA Fusion Protein; Drug: Vincristine Liposomal

INTERVENTIONS:
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
  Arms: Arm A (sEPHB4-HSA, cytarabine)
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Recombinant EphB4-HSA Fusion Protein — Given IV
  Other Names: sEphB4-HSA
Drug: Vincristine Liposomal — Given IV
  Other Names: Lipid-Encapsulated Vincristine; Liposomal Vincristine; Onco TCS; Vincacine; VincaXome; Vincristine Liposome; Vincristine, Liposomal
  Arms: Arm B (sEPHB4-HSA, vincristine liposomal)

SUMMARY:
This phase I trial studies the side effects and best dose of recombinant EphB4-HSA fusion protein when given together with cytarabine or vincristine liposomal in treating participants with acute leukemia that has come back or has not responded to treatment. Drugs used in chemotherapy, such as recombinant ephb4-HSA fusion protein, cytarabine, and vincristine liposomal, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving the drugs in different combinations may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Characterize the DLTs (dose limiting toxicities) and overall toxicity profile of recombinant EphB4-HSA fusion protein (sEPHB4-HSA) as a single agent and in combination with cytarabine or liposomal vincristine in patients with acute leukemia.

SECONDARY OBJECTIVES:

I. Estimate the clinical response (including minimal residual disease [MRD]) in blood and bone marrow of sEPHB4-HSA in combination with cytarabine in patients with relapsed/refractory acute myeloid leukemia.

II. Estimate the clinical response (including MRD) in blood and bone marrow of sEPHB4-HSA in combination with liposomal vincristine in patients with relapsed/refractory acute lymphoid leukemia.

III. Estimate the single agent clinical response of sEPHB4-HSA in blood and bone marrow of patients with relapsed/refractory acute myeloid leukemia (AML) or acute lymphoid leukemia (ALL).

IV. Assess pharmacokinetics of sEPHB4-HSA as a single agent and in combination with cytarabine or liposomal vincristine in patients with leukemia.

EXPLORATORY OBJECTIVES:

I. Estimate progression-free survival and overall survival in patients treated with sEPHB4-HSA in combination with cytarabine or liposomal vincristine.

II. Estimate percentage of patients proceeding to allogeneic stem cell transplantation.

III. Correlate expression of EPHB4 leukemic blasts and ephrinB2 in bone marrow microenvironment with response to sEPHB4-HSA.

IV. Evaluate the effect of sEPHB4-HSA on downstream protein mediators of the EPHB4 pathway (phosphorylated [p]AKT, pS6) on leukemic blasts and determine if these can be used as biomarkers of response to treatment.

V. Profile the immuno-modulatory effects of sEPHB4-HSA on peripheral blood leukocytes and in the tumor microenvironment.

OUTLINE: This is a dose-escalation study of recombinant EphB4-HSA fusion protein. Participants are randomized to 1 of 2 arms.

ARM A: Participants receive recombinant EphB4-HSA fusion protein intravenously (IV) over 60 minutes on days 1, 8, 15, and 22 and cytarabine IV over 4 hours on days 1-5. Treatment repeats every 28 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.

ARM B: Participants receive recombinant EphB4-HSA fusion protein IV over 60 minutes on days 1, 8, 15, and 22 and vincristine liposomal IV over 60 minutes on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of relapsed or refractory acute leukemia (acute myeloid leukemia, acute lymphoblastic leukemia, blast crisis of chronic myeloid leukemia [CML], secondary AML from prior myelodysplastic syndrome [MDS] / myeloproliferative neoplasm [MPN]); minimum of 5% blasts in the bone marrow or 10% blasts in circulation
* Patients with Philadelphia chromosome (Ph)+ ALL or blast crisis of CML must be refractory (not intolerant) to at least 2 second/third generation ABL kinase inhibitors (TKI)
* For AML: patients must belong to one of the following ?high risk? categories:

  * Primary induction failure (PIF) as defined by failure to achieve at least a 50% reduction in bone marrow blasts after one cycle of high intensity, anthracycline containing induction regimen or failure to achieve complete response (CR)/complete remission with incomplete blood count recovery (CRi) after two cycles of high intensity chemotherapy
  * First early relapse as defined by an initial remission duration of fewer than 6 months
  * Second or subsequent relapse regardless of remission duration, or
  * Relapse after allogeneic or autologous stem cell transplantation (first relapse after stem cell transplant would be eligible, regardless of prior duration of remission)
* Patients with MDS who transform to AML while on hypomethylator agents or patients with AML who progress on hypomethylator agents could be considered for arm A of this trial if

  * They choose not to be treated on or are ineligible for the investigator's competing trial of sEPHB4-HSA + hypomethylator (9L-16-6)
  * They are appropriate for high dose cytarabine treatment
* For ALL: patients must belong to one of the following ?high risk? categories:

  * Primary refractory as defined by failure to achieve CR after induction and at least one salvage therapy
  * Second or subsequent relapse
  * Relapse after allogeneic or autologous stem cell transplantation (requirement for second relapse does not apply post-transplant)
  * All variants of ALL including T-ALL, B / myeloid, lymphoblastic leukemia lymphoma are eligible
* Patients with myeloid diseases (AML, myeloid blast crisis of CML) will be eligible for arm A with cytarabine; patients with lymphoid diseases (ALL, lymphoid blast crisis of CML) will be eligible for arm B with liposomal vincristine; patients with leukemia of ambiguous lineage or bi-phenotypic leukemia (e.g. B/myeloid) may be treated on either arm A or B, at discretion of treating physician
* Performance status Eastern Cooperative Oncology Group (ECOG) 0 to 2
* Life expectancy > 2 months
* Total bilirubin ? 3 X upper limit of normal (ULN), unless attributable to Gilbert syndrome
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) / alanine transaminase [ALT] (serum glutamic pyruvic transaminase [SPGT]) ? 5 X institutional upper limit of normal
* Creatinine: glomerular filtration rate (GFR) > 30 as calculated by modification of diet in renal disease (MDRD) equation
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* No major surgery within 4 weeks of first dose of sEPHB4
* Peripheral blood blast count ? 30,000 at time of eligibility assessment (within 7 days of start of therapy); blast counts that increase beyond 30,000 after a patient is deemed eligible will not disqualify the patient
* For subjects with prior allogeneic stem cell transplant, no evidence of active graft-versus host disease (GVHD), and must be ? 2 weeks off immunosuppressive therapy
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Diagnosis of acute promyelocytic leukemia (M3 classification)
* ALL patient refractory to their first induction only or their first relapse, will be excluded; they must be refractory to at least one salvage therapy, or relapse after first salvage, to be eligible
* ALL patients refractory to liposomal vincristine as defined by progression while on therapy or relapse within 3 months of completion of therapy with liposomal vincristine
* Prior malignancy requiring therapy within the last 12 months (excluding non-melanoma skin cancer); hormone therapy for prostate cancer or adjuvant endocrine therapy for breast cancer would not be excluded
* Patient is receiving other investigational agents
* Active central nervous system (CNS) disease

  * Definition: any patient receiving active CNS therapy (defined as more than 1 intrathecal treatment per week or current radiation therapy to brain); if patient has a history of CNS disease: must have cerebrospinal fluid (CSF) sampling within 28 days of enrollment that is negative for leukemia; intrathecal chemotherapy for patients without active CNS disease is allowed (e.g., ongoing primary or secondary prophylaxis for patients who cleared the CSF prior to study enrollment); CSF sample is not required for enrollment for patients with no history of CNS disease
* Chemotherapy within 2 weeks of first dose of sEPHB4-HSA (minimum of 6 weeks for nitrosoureas and 8 weeks for bone marrow transplantation) with the following exceptions:

  * Hydroxyurea allowed prior to, and up to day +5 of cycle 0 of treatment (max 100 mg/kg/day)
  * Corticosteroids allowed until day -3 (max dexamethasone 20mg/day)
  * Maintenance chemotherapy for ALL allowed one week prior to start of treatment (e.g., POMP)
* Grade ? 2 toxicity (other than alopecia) continuing from prior anticancer therapy, including radiation
* Patients with Charcot-Marie-Tooth disease or other demyelinating diseases are excluded from the liposomal vincristine containing arm
* New York Heart Association class 3 or 4 heart failure; myocardial infarction, acute coronary syndrome, diabetes mellitus with ketoacidosis, or chronic obstructive pulmonary disease (COPD) requiring hospitalization in the preceding 6 months; or any other intercurrent medical condition that contraindicates treatment with sEPHB4-HSA or places the patient at undue risk for treatment related complications
* Uncontrolled active systemic infections
* Known history of human immunodeficiency virus (HIV) or active infection with hepatitis C virus (HCV) or hepatitis B virus (HBV); patients with HBV and/or HCV sero-positivity only will be eligible, if nucleic acid amplification testing (NAT) is negative
* Warfarin (any dose) or full-dose anticoagulation with other agents (low molecular weight heparin, antithrombin agents, anti-platelet agents and full dose aspirin) within 7 days prior to first dose of study drug; patients on prophylactic doses of low-molecular weight heparin are allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2020-11-24 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 24 months
  Will be assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.03 and summarized for each course separately.
Best clinical response in the blood and bone marrow observed at anytime during single agent treatment with recombinant EphB4-HSA fusion protein alone | Up to 24 months
  Best clinical response defined as complete remission (CR) + complete remission with incomplete blood count recovery (CRi) + partial remission (PR) + partial remission with incomplete blood count recovery (PRi).
  CR defined as Neutrophils: >1,000/µL; Platelets: >100,000/µL; Bone Marrow Blasts: <5% with spicules, no Auer rods; Other: Transfusion independent, no extra medullary disease.
  CRi defined as Neutrophils: <1,000/µL; Platelets: <100,000/µL; Bone Marrow Blasts: <5%; Other: Either neutrophils or platelets not recovered, no extra medullary disease.
  PR defined as Neutrophils: >1,000/µL; Platelets: >100,000/µL; Bone Marrow Blasts: decrease to 5-25 and = > 50% decrease from start.
  PRi defined as Neutrophils: <1,000/µL; Platelets: <100,000/µL; Bone Marrow Blasts: decrease to 5-25 and = > 50% decrease from start.
Complete remission (CR) and complete remission with incomplete blood count recovery (CRi) observed at anytime for the combination with cytarabine or liposomal vincristine | Up to 24 months
  CR defined as Neutrophils: >1,000/µL; Platelets: >100,000/µL; Bone Marrow Blasts: <5% with spicules, no Auer rods; Other: Transfusion independent, no extra medullary disease.
  CRi defined as Neutrophils: <1,000/µL; Platelets: <100,000/µL; Bone Marrow Blasts: <5%; Other: Either neutrophils or platelets not recovered, no extra medullary disease.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 24 months
  Will be calculated for all patients who achieve a CR or CRi from first documentation ofCR or CRi to recurrence or death.

CONTACTS AND LOCATIONS:
Overall Officials: Akil Merchant, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States